CLINICAL TRIAL: NCT02509546
Title: A Phase I/II Trial of 8-Chloro-Adenosine in Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: 8-Chloroadenosine in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 14269; NCI-2015-00871 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 123456; 122489; 14269 (Other: City of Hope Comprehensive Cancer Center)
Record Dates: First submitted 2015-06-10; First posted 2015-07-28 (Estimated); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Acute Myeloid Leukemia Arising From Previous Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — 8-chloroadenosine; beta-apocarotenoid-14',13'-dioxygenase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Phase I - 100mg/m^2 1-hour infusion (Experimental): 100mg/m^2 8-chloro-adenosine administered a one-hour intravenous infusion daily for first 5 days of each 28-day cycle, up to four cycles.
  Interventions: Drug: 8-Chloroadenosine; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Phase I - 200mg/m^2 1-hour infusion (Experimental): 200mg/m^2 8-chloro-adenosine administered a one-hour intravenous infusion daily for first 5 days of each 28-day cycle, up to four cycles.
  Interventions: Drug: 8-Chloroadenosine; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Phase I - 400mg/m^2 1-hour infusion (Experimental): 400mg/m^2 8-chloro-adenosine administered a one-hour intravenous infusion daily for first 5 days of each 28-day cycle, up to four cycles.
  Interventions: Drug: 8-Chloroadenosine; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Phase I - 800mg/m^2 1-hour infusion (Experimental): 800mg/m^2 8-chloro-adenosine administered a one-hour intravenous infusion daily for first 5 days of each 28-day cycle, up to four cycles.
  Interventions: Drug: 8-Chloroadenosine; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Phase I - 400mg/m^2 4-hour infusion (Experimental): 400mg/m^2 8-chloro-adenosine administered a four-hour intravenous infusion daily for first 5 days of each 28-day cycle, up to four cycles.
  Interventions: Drug: 8-Chloroadenosine; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study
- Phase I - 600mg/m^2 4-hour infusion (Experimental): 600mg/m^2 8-chloro-adenosine administered a four-hour intravenous infusion daily for first 5 days of each 28-day cycle, up to four cycles.
  Interventions: Drug: 8-Chloroadenosine; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study

INTERVENTIONS:
Drug: 8-Chloroadenosine — Given IV
  Other Names: 8-Chloro-adenosine; 8-Cl-adenosine; 8-Cl-Ado
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase I/II trial studies the side effects and best dose of 8-chloroadenosine and to see how well it works in treating patients with acute myeloid leukemia that has returned after a period of improvement (relapsed) or does not respond to treatment (refractory). Drugs used in chemotherapy, such as 8-chloroadenosine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the maximum tolerated dose (recommended phase II dose, RP2D) of 8-chloro-adenosine, when given as a single agent, in patients with relapsed or refractory acute myeloid leukemia. (Phase I) II. To assess tolerability and safety of 8-chloro-adenosine at each dose level by evaluation of toxicities including: type, frequency, severity, attribution, time course and duration. (Phase I) III. To estimate the response rate and to evaluate the antitumor activity of 8-chloro-adenosine, when given as a single agent, as assessed by complete remission rate (complete remission [CR] + complete remission with incomplete blood count recovery [CRi]). (Phase II)

SECONDARY OBJECTIVES:

I. To evaluate for disease response to 8-chloro-adenosine in refractory/relapsed acute myeloid leukemia (AML) on each dose level tested. (Phase I) II. To obtain estimates of remission duration and survival probabilities (overall and event-free). (Phase II) III. To obtain an estimate of the overall response rate (CR + CRi + partial response [PR]). (Phase II) IV. To summarize and evaluate toxicities by type, frequency, severity, attribution, time course and duration. (Phase II)

CLINICAL PHARMACOLOGY OBJECTIVES:

I. To describe the plasma, urinary and cellular pharmacokinetics of 8-chloro-adenosine and metabolites.

II. To determine the impact of 8-chloro-adenosine on cellular adenosine triphosphate (ATP) pool in AML blasts.

III. To assess the impact of 8-chloro-adenosine therapy on select short-lived messenger (m) ribonucleic acids (RNAs) and corresponding proteins in circulating AML blasts.

IV. To correlate clinical responses and toxicity with plasma/urine 8-chloro-adenosine level (pharmacokinetic [PK]), cellular 8-chloro-ATP (PK) and cellular ATP pool.

EXPLORATORY EX-VIVO MOLECULAR OBJECTIVES:

I. To determine the cytotoxicity of 8-chloro-adenosine toward leukemic progenitor cells in vitro.

II. To generate a preliminary pre-treatment RNA/micro RNA (miRNA) signature in leukemic progenitor cells, and explore its possible association with in vitro cytotoxicity to 8-chloro-adenosine.

III. To explore the possible association between the preliminary RNA/miRNA signature and clinical response to 8-chloro-adenosine.

OUTLINE: This is a phase I, dose-escalation study followed by a phase II study.

Patients receive 8-chloro-adenosine intravenously (IV) over 4 hours on days 1-5. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and then every 3 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must have the ability to understand and the willingness to sign a written informed consent
* Patients must have a life expectancy of > 3 months
* Patients must exhibit an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2
* Patients must have a diagnosis of AML as per World Health Organization (WHO) Classification of Hematologic Neoplasms
* Patients must meet one of the three treatment history criteria:

  * Relapsed AML who have failed at least 1 line of salvage therapy
  * De novo AML who have not achieved CR after 2 lines of therapy
  * AML evolving from myelodysplastic syndrome (MDS) or myeloproliferative disorder who have failed hypomethylating agent or induction chemotherapy
  * Patients who have relapsed after allogeneic hematopoietic cell transplant (HCT) are eligible if they are at least 3 months after HCT, do not have active graft vs. host disease (GVHD) and are off immunosuppression except for maintenance dose of steroids (prednisone 10 mg/day or less)
* At least 2 weeks from prior chemotherapy or radiation therapy to time of start of treatment, except for hydroxyurea or corticosteroid therapy which may be continued through cycle 1
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 2.5 x upper limit of normal (ULN)
* Total bilirubin =< 1.5 X ULN
* Corrected QT (QTc) =< 480 ms
* Calculated creatinine clearance (CrCl) >= 50 mL/min per 24 hour urine collection or the Cockcroft-Gault formula
* Negative serum or urine beta-human chorionic gonadotropin (beta-HCG) test (female of childbearing potential only), to be performed locally within the screening period
* Agreement by females of childbearing potential and sexually active males to use an effective method of contraception (hormonal or barrier method of birth control or abstinence) prior to study entry and for three months following duration of study participation; the effects of study treatment on a developing fetus have the potential for teratogenic or abortifacient effects; should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately

Exclusion Criteria:

* Current or planned use of other investigational agents, or concurrent biological chemotherapy, or radiation therapy during the study treatment period
* Expected to undergo HCT within 120 days of enrollment
* Current or planned use of agents that prolong or suspected to prolong QTc
* Diagnosis of acute promyelocytic leukemia
* Active central nervous system leukemia
* Active fungal infection or bacterial sepsis
* Active peptic ulcer disease
* History of heart failure or cardiac arrhythmia
* Other active malignancy except for localized skin cancer, bladder, prostate, breast or cervical carcinoma in situ
* Pregnant women and women who are lactating; 8-chloro-adenosine is an agent with the potential for teratogenic or abortifacient effects; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with 8-chloro-adenosine, breastfeeding should be discontinued if the mother is treated with 8-chloro-adenosine
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-09-02 (Actual); Primary Completion 2021-03-09 (Actual); Study Completion 2021-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vinod Pullarkat, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The phase 2 portion was not pursued since no marrow complete remissions were observed with single agent therapy and a decision was made to pursue a combination trial with the Bcl-2 inhibitor venetoclax based on preclinical data.
Period: Overall Study
Arm/Group | Phase I - 100mg/m^2 1-hour Infusion | Phase I - 200mg/m^2 1-hour Infusion | Phase I - 400mg/m^2 1-hour Infusion | Phase I - 800mg/m^2 1-hour Infusion | Phase I - 400mg/m^2 4-hour Infusion | Phase I - 600mg/m^2 4-hour Infusion
Started | 3 | 3 | 4 | 2 | 2 | 6
Completed | 3 | 3 | 4 | 2 | 2 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I - 100mg/m^2 8-chloro-adenosine 1-hour Infusion: 100mg/m^2 8-chloro-adenosine administered a one-hour intravenous infusion daily for first 5 days of each 28-day cycle, up to four cycles.
- Phase I - 200mg/m^2 8-chloro-adenosine 1-hour Infusion: 200mg/m^2 8-chloro-adenosine administered a one-hour intravenous infusion daily for first 5 days of each 28-day cycle, up to four cycles.
- Phase I - 400mg/m^2 8-chloro-adenosine 1-hour Infusion: 400mg/m^2 8-chloro-adenosine administered a one-hour intravenous infusion daily for first 5 days of each 28-day cycle, up to four cycles.
- Phase I - 800mg/m^2 8-chloro-adenosine 1-hour Infusion: 800mg/m^2 8-chloro-adenosine administered a one-hour intravenous infusion daily for first 5 days of each 28-day cycle, up to four cycles.
- Phase I - 400mg/m^2 8-chloro-adenosine 4-hour Infusion: 400mg/m^2 8-chloro-adenosine administered a four-hour intravenous infusion daily for first 5 days of each 28-day cycle, up to four cycles.
- Phase I - 600mg/m^2 8-chloro-adenosine 4-hour Infusion: 600mg/m^2 8-chloro-adenosine administered a four-hour intravenous infusion daily for first 5 days of each 28-day cycle, up to four cycles.
- Total: Total of all reporting groups
Arm/Group | Phase I - 100mg/m^2 8-chloro-adenosine 1-hour Infusion | Phase I - 200mg/m^2 8-chloro-adenosine 1-hour Infusion | Phase I - 400mg/m^2 8-chloro-adenosine 1-hour Infusion | Phase I - 800mg/m^2 8-chloro-adenosine 1-hour Infusion | Phase I - 400mg/m^2 8-chloro-adenosine 4-hour Infusion | Phase I - 600mg/m^2 8-chloro-adenosine 4-hour Infusion | Total
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 2 | 6 | 20
Age, Continuous [Median (Full Range); unit: years] | 75 [69 to 77] | 54 [28 to 66] | 59 [45 to 71] | 56 [50 to 63] | 68 [59 to 77] | 70 [61 to 75] | 66 [28 to 77]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 2 | 1 | 4 | 12
  Male | 2 | 2 | 1 | 0 | 1 | 2 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 1 | 1 | 0 | 3 | 7
  Not Hispanic or Latino | 3 | 1 | 3 | 1 | 2 | 3 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 4 | 2 | 2 | 6 | 20

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Dose (RP2D) of 8-Chloro-adenosine (8-Cl-Ado)
Description: According to the standard 3+3 rules, where the highest DL that produced ≤ 1/6 DLTs in cycle 1 would be defined as the maximum tolerated dose (MTD). The RP2D of 8-Cl-Ado would generally be the MTD, but it could be less than the initially calculated MTD as determined from a review of the available data and cumulative toxicities from phase 1.
Time Frame: Up to 28 days following first study agent administration.
Population: 3 patients at 100 mg/m^2 1-hr; 3 patients at 200 mg/m^2 1-hr; 4 patients at 400 mg/m^2 1-hr; 2 patients at 800 mg/m^2 1-hr; 2 patients at 400 mg/m^2 4-hr; 6 patients at 600 mg/m^2 4-hr.
Measure: Number; unit: mg/m^2
Groups:
- Phase I - Treatment (8-chloro-adenosine): Patients receive 8-chloro-adenosine IV on days 1-5. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.
Arm/Group | Phase I - Treatment (8-chloro-adenosine)
Number analyzed (Participants) | 20
mg/m^2 | 400

2. Primary Outcome: Dose Limiting Toxicity (DLT)
Description: Toxicity was graded according to the NCI-Common Terminology Criteria for Adverse Events version 4.03. A DLT was defined as any of the following toxicities (please see the details in section of 13.2 of the protocol) that occur during cycle 1, per CTCAE version 4.03, and were considered related to the study drug.
Time Frame: Up to 28 days following first study agent administration.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I - 100mg/m^2 8-chloro-adenosine 1-hour Infusion | Phase I - 200mg/m^2 8-chloro-adenosine 1-hour Infusion | Phase I - 400mg/m^2 8-chloro-adenosine 1-hour Infusion | Phase I - 800mg/m^2 8-chloro-adenosine 1-hour Infusion | Phase I - 400mg/m^2 8-chloro-adenosine 4-hour Infusion | Phase I - 600mg/m^2 8-chloro-adenosine 4-hour Infusion
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 2 | 6
Participants | 0 | 0 | 1 | 2 | 0 | 2

3. Secondary Outcome: Complete Remission Rate (CR + CRi)
Description: Complete remission rate (CR + CRi) based on the Döhner 2010 criteria and calculated as the percent of evaluable patients that have confirmed CR or CRi is to evaluate the antitumor activity of 8-chloro-adenosine.
Time Frame: Up to 2 years following first study agent administration.
Measure: Number; unit: Percent of evaluable patients
Arm/Group | Phase I - 100mg/m^2 8-chloro-adenosine 1-hour Infusion | Phase I - 200mg/m^2 8-chloro-adenosine 1-hour Infusion | Phase I - 400mg/m^2 8-chloro-adenosine 1-hour Infusion | Phase I - 800mg/m^2 8-chloro-adenosine 1-hour Infusion | Phase I - 400mg/m^2 8-chloro-adenosine 4-hour Infusion | Phase I - 600mg/m^2 8-chloro-adenosine 4-hour Infusion
Number analyzed (Participants) | 3 | 3 | 4 | 2 | 2 | 6
Percent of evaluable patients | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 2 years following first study agent administration.
Arm/Group | Phase I - 100mg/m^2 8-chloro-adenosine 1-hour Infusion | Phase I - 200mg/m^2 8-chloro-adenosine 1-hour Infusion | Phase I - 400mg/m^2 8-chloro-adenosine 1-hour Infusion | Phase I - 800mg/m^2 8-chloro-adenosine 1-hour Infusion | Phase I - 400mg/m^2 8-chloro-adenosine 4-hour Infusion | Phase I - 600mg/m^2 8-chloro-adenosine 4-hour Infusion
All-Cause Mortality (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 2/2 | 2/2 | 6/6
Serious Adverse Events (participants affected / at risk) | 1/3 | 1/3 | 2/4 | 2/2 | 2/2 | 6/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 4/4 | 2/2 | 2/2 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - 100mg/m^2 8-chloro-adenosine 1-hour Infusion (N=3) | Phase I - 200mg/m^2 8-chloro-adenosine 1-hour Infusion (N=3) | Phase I - 400mg/m^2 8-chloro-adenosine 1-hour Infusion (N=4) | Phase I - 800mg/m^2 8-chloro-adenosine 1-hour Infusion (N=2) | Phase I - 400mg/m^2 8-chloro-adenosine 4-hour Infusion (N=2) | Phase I - 600mg/m^2 8-chloro-adenosine 4-hour Infusion (N=6)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MULTIORGAN FAILURE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ASPERGUILLUS GALACTOMANNAN (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
LUNG INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
DISEASE PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LEUKEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INVASIVE PULMONARY ASPERGILLOSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I - 100mg/m^2 8-chloro-adenosine 1-hour Infusion (N=3) | Phase I - 200mg/m^2 8-chloro-adenosine 1-hour Infusion (N=3) | Phase I - 400mg/m^2 8-chloro-adenosine 1-hour Infusion (N=4) | Phase I - 800mg/m^2 8-chloro-adenosine 1-hour Infusion (N=2) | Phase I - 400mg/m^2 8-chloro-adenosine 4-hour Infusion (N=2) | Phase I - 600mg/m^2 8-chloro-adenosine 4-hour Infusion (N=6)
ANEMIA (Blood and lymphatic system disorders) | 3 (33) | 3 (46) | 3 (31) | 1 (16) | 2 (20) | 6 (48)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 2 (2) | 1 (6) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LYMPH NODE PAIN (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ATRIAL ARRHYTHMIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (5) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
ATRIAL FLUTTER (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARDIAC ARREST (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
CARDIOMEGALY (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CHEST PAIN CARDIAC (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DILATED CARDIOMYOPATHY (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEART FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
MYOCARDITIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PAROXYSMAL ATRIAL TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PERICARDIAL EFFUSION (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SINUS BRADYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1) | 3 (17) | 3 (5) | 1 (1) | 0 (0) | 6 (17)
SUPERVENTRICULAR SINUS TACYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
T WAVE CHANGES (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VENTRICULAR FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
DRY EYE (Eye disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
EYE PAIN (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
WATERING EYES (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 2 (4) | 3 (5) | 1 (1) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (2)
BLOATING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
CONSTIPATION (Gastrointestinal disorders) | 2 (2) | 1 (2) | 1 (5) | 1 (1) | 1 (1) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 2 (5) | 3 (7) | 2 (3) | 0 (0) | 0 (0) | 3 (6)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 2 (2)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
ENTEROCOLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FECAL INCONTINENCE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GERD (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GINGIVAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
HEMORRHOIDS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LOWER GASTROINTESTINAL HEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 1 (6) | 2 (6) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 1 (1) | 2 (10) | 3 (7) | 2 (6) | 1 (1) | 4 (9)
ORAL PAIN (Gastrointestinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 1 (1) | 2 (9) | 2 (4) | 1 (3) | 0 (0) | 4 (15)
CHILLS (General disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1)
DIAPHORESIS (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
EDEMA FACE (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
EDEMA LIMBS (General disorders) | 2 (2) | 2 (4) | 2 (3) | 1 (1) | 0 (0) | 4 (8)
FACIAL PAIN (General disorders) | 0 (0) | 1 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
FATIGUE (General disorders) | 1 (2) | 1 (2) | 2 (3) | 1 (22) | 2 (3) | 4 (6)
FEVER (General disorders) | 0 (0) | 1 (7) | 4 (10) | 2 (7) | 0 (0) | 3 (6)
FLUID OVERLOAD (General disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFUSION SITE EXTRAVASATION (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LOCALIZED EDEMA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 3 (3)
MALAISE (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MULTIORGAN FAILURE (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
NONCARDIAC CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 2 (2)
PAIN (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
PAIN AT IV SITE (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALLERGIC REACTION (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
C. DIFFICILE COLITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CATHETER RELATED INFECTION (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LUNG INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BRUISING (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4)
VASCULAR ACCESS COMPLICATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
ACTIVATED PARTIAL THROMBOPLASTIN TIME PROLONGED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 3 (3)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1) | 2 (5) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (6)
BLOOD BILIRUBIN INCREASED (Investigations) | 3 (8) | 3 (12) | 2 (5) | 2 (4) | 2 (3) | 6 (17)
CARDIAC TROPONIN I INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CARDIAC TROPONIN T INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CPK INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CREATININE INCREASED (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (7)
EJECTION FRACTION DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ELECTROCARDIOGRAM QT CORRECTED INTERVAL PROLONGED (Investigations) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 5 (23)
LYMPHOCYTE COUNT DECREASED (Investigations) | 2 (9) | 3 (21) | 2 (17) | 1 (10) | 2 (3) | 5 (11)
LYMPHOCYTE COUNT INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (10) | 0 (0) | 2 (6) | 0 (0) | 2 (8) | 5 (30)
PLATELET COUNT DECREASED (Investigations) | 3 (59) | 3 (52) | 3 (6) | 1 (1) | 2 (25) | 5 (36)
WEIGHT GAIN (Investigations) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WEIGHT LOSS (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 5 (16)
WHITE BLOOD CELL DECREASED (Investigations) | 3 (13) | 2 (10) | 2 (6) | 1 (5) | 2 (6) | 5 (20)
ACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
ALKALOSIS (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
ANOREXIA (Metabolism and nutrition disorders) | 2 (2) | 3 (6) | 3 (4) | 1 (1) | 2 (2) | 5 (5)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (10) | 1 (1) | 0 (0) | 0 (0) | 1 (7) | 1 (1)
HYPERKALEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERMAGNESEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (5)
HYPERNATREMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
HYPERTRIGLYCERIDEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 3 (12) | 3 (15) | 4 (10) | 1 (1) | 1 (2) | 6 (19)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 3 (10) | 1 (3) | 1 (1) | 2 (5) | 0 (0) | 2 (4)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
HYPOKALEMIA (Metabolism and nutrition disorders) | 2 (13) | 3 (12) | 4 (10) | 2 (15) | 0 (0) | 6 (28)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 2 (7) | 2 (3) | 2 (3) | 1 (2) | 0 (0) | 4 (11)
HYPONATREMIA (Metabolism and nutrition disorders) | 3 (14) | 3 (8) | 3 (6) | 1 (10) | 1 (1) | 5 (17)
HYPOPHOSPHATEMIA (Metabolism and nutrition disorders) | 2 (5) | 2 (3) | 3 (9) | 2 (14) | 1 (2) | 5 (12)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3) | 1 (1) | 2 (3) | 1 (1) | 2 (4)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 1 (2)
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
GENERALIZED MUSCLE WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 5 (8)
JOINT RANGE OF MOTION DECREASED (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (3)
LEFT SCAPULA PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3)
RIGHT SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE MYELOGENOUS LEUKEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE MYELOID LEUKEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DISEASE PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
REFRACTORY RELAPSED ACUTE MYELOID LEUKEMIA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (3)
DYSARTHRIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (3) | 2 (8) | 1 (4) | 0 (0) | 0 (0) | 2 (3)
LETHARGY (Nervous system disorders) | 1 (3) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
MEMORY IMPAIRMENT (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
PRESYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SOMNOLENCE (Nervous system disorders) | 1 (1) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TREMOR (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
AGITATION (Psychiatric disorders) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (4)
ANXIETY (Psychiatric disorders) | 1 (1) | 1 (6) | 2 (3) | 1 (1) | 0 (0) | 3 (6)
CONFUSION (Psychiatric disorders) | 1 (4) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
DELIRIUM (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INSOMNIA (Psychiatric disorders) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 4 (5)
RESTLESSNESS (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FLUID RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEMATURIA (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 2 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GENITAL EDEMA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PERINEAL PAIN (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SCROTAL EDEMA (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VAGINAL HEMORRHAGE (Reproductive system and breast disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALLERGIC RHINITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ATELECTASIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
BRONCHOPULMONARY HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (6) | 2 (2) | 1 (1) | 0 (0) | 2 (3)
DECREASED FEV (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 2 (3) | 4 (6) | 0 (0) | 0 (0) | 4 (8)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 3 (5)
FUNGAL SINUSITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GENERALIZED EDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (11)
LARYNGEAL HEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
LARYNGEAL INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LIGHT GRAM POSITIVE COCCI (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LUNG INFILTRATES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NASAL CONGESTION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1)
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PULMONARY INFILTRATES (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
RHINITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RHINORRHEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
RUNNY NOSE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SORE THROAT (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 1 (3) | 0 (0) | 0 (0) | 3 (3)
TACHYPNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4)
VOICE ALTERATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
WHEEZING (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALOPECIA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
BLISTER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIAPHORESIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
ERYTHEMATOUS FOLLICULAR RASH (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PALMARPLANTAR ERYTHRODYSESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PERIORBITAL EDEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
PETICHIAE (CHEST) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKIN DISCOLORATION (HANDS) (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKIN DISCOLORATION FEET (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKIN HYPERPIGMENTATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HICKMAN SITE DISCOMFORT (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLUSHING (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEMATOMAS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 3 (23) | 3 (21) | 4 (9) | 2 (10) | 2 (18) | 6 (31)
HYPOTENSION (Vascular disorders) | 2 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (6)
SUPERFICIAL THROMBOPHLEBITIS (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/46/NCT02509546/Prot_SAP_000.pdf